CLINICAL TRIAL: NCT04310839
Title: Outpatient Management of Patients With a Left Laparoscopic Colectomy
Brief Title: Outpatient Left Laparoscopic Colectomy
Acronym: COATI
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de la Rochelle Ré Aunis (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018/P01/280
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Colonic Neoplasms; Colonic Diverticulosis
MeSH Terms: conditions — Colonic Neoplasms; Diverticulosis, Colonic | interventions — Colectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- outpatient left laparoscopic colectomy: Left laparoscopic laparoscopic colectomy patient managed on an outpatient basis
  Interventions: Procedure: Colectomy

INTERVENTIONS:
Procedure: Colectomy — colectomy due to neoplastic (stage 1) or diverticulosis

SUMMARY:
The success of the enhanced recovery program after surgery leads us to consider outpatient management of the colectomy. To this end, the investigators have designed an observational and prospective study of left laparoscopic colectomy on an outpatient basis. The objective is to assess the harmlessness of this management compared to standard management in the context of a public hospital.

DETAILED DESCRIPTION:
In France, colectomy represents about 40,000 interventions per year, most of them scheduled, and 2/3 in a context of neoplasia. This surgery is associated with numerous postoperative complications. Since the start of Enhanced Recovery After Surgery (ERAS) in 1997, complications have been steadily reduced by optimizing surgical and anaesthetic techniques. At the same time, the average length of post-operative stay has decreased. In 2014, ERAS was the subject of recommendations by the French Society of Anaesthesia and Resuscitation, taken up by the French Health Authority (HAS) in 2016, and which are now an integral part of surgical management in colorectal surgery. More recently, two teams have set up an outpatient colectomy program. The three studies published on this subject show encouraging results, in a private structure, with no increase in postoperative complications.

In accordance with the recommendations on ERAS published by the HAS, a program involving pre-, per- and post-interventional investment, has been put in place. Patients are discharged on D0, followed by close monitoring by a home care nurse twice daily. This nurse is in charge of collecting clinical data in order to detect possible early signs of post-operative complications that would justify re-hospitalisation after a medical-surgical decision.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Classification (ASA) score I and II,
* Patient with an indication for scheduled left colectomy due to neoplastic (stage 1) or diverticulitis,
* Patient residing less than 30 minutes from La Rochelle hospital,
* Presence of a companion from the anaesthesia consultation onwards,
* Presence of an attendant at the patient's discharge,
* Perfect understanding of outpatient care, pathology and surgical procedure of the patient and accompanying person,
* Informed of the study.

Exclusion Criteria:

* ASA score 3 et 4,
* Indication for a straight or transverse colectomy,
* Neoplasia evolution > stage 1,
* Presence of anticoagulant treatment,
* Intraoperative bleeding > 500ml,
* Conversion to laparotomy,
* Severe anesthetic complication (Anaphylaxis, Difficult Intubation),
* Persons deprived of their liberty by a judicial or administrative decision,
* Persons of full age who are subject to a legal protection measure,
* Persons unable to consent,
* Persons who are not members of or beneficiaries of a social security scheme,
* Patient's refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients taken care for a left colectomy due to colonic neoplasm or diverticulosis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
30-day readmission rate | 30 days after surgery
  Number of re-hospitalisation after a medical-surgical decision due to post-operative complications

SECONDARY OUTCOMES:
Pain measurement: pain rating scale | 7 days after surgery
  Score at the numerical pain rating scale
Mobilization | Day 0
  Time (in hours) between extubation and first mobilization
Ileus | up to 7 days after surgery
  Number of day between surgery and first gas / stool

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Smirnoff, MD, Study Director — Groupe Hospitalier de la Rochelle Ré Aunis
Locations (1):
- Groupe Hospitalier de la Rochelle Ré Aunis, La Rochelle, France

IPD SHARING:
Plan to Share IPD: Undecided